CLINICAL TRIAL: NCT06688526
Title: Auditory Stimulation Effect on Brain Oscillations and Sleep Dependent Learning
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Catherine Chu, MD, Associate Professor, Neurology, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2024P002714
Record Dates: First submitted 2024-10-25; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Healthy Control

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Auditory Stimulation (Active Comparator): Quiet sounds are played during sleep
  Interventions: Other: Quiet Sounds
- Sham Stimulation (Sham Comparator): Volume is set to zero.
  Interventions: Other: Sham sounds

INTERVENTIONS:
Other: Quiet Sounds — Quiet sounds are played during sleep
  Arms: Auditory Stimulation
Other: Sham sounds — No sounds are played during sleep
  Arms: Sham Stimulation

SUMMARY:
The investigators are testing the impact of quiet sounds played during sleep on brain oscillations and memory.

DETAILED DESCRIPTION:
Participants will undergo two visits with a memory task and nap. During one of the visits, quiet sounds will be played timed with sleep oscillations. During the other visit, no sounds will be played. Brain oscillations and memory will be measured at each visit.

ELIGIBILITY:
Inclusion Criteria: Adult -

Exclusion Criteria: History of neurological disease, psychiatric disease, sleep apnea or sleep disorder.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-13 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Sleep spindle rate | 90 minutes
  Sleep spindles are prominent thalamocortical brain oscillations seen on EEG during sleep that have been mechanistically linked to sleep-dependent memory consolidation. The sleep spindle rate over the course of the nap will be assessed using an automated spindle detector applied to the collected EEG sleep data.

SECONDARY OUTCOMES:
Memory consolidation | 90 minutes
  The motor sequence task (MST), a validated probe of memory consolidation, will be used to measure sleep-dependent memory consolidation. Participants will trained on MST before the nap opportunity and tested on MST after the nap opportunity to reliably measure memory consolidation.

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared upon request to the study PI
Time Frame: within one year of study termination
Access Criteria: Academic investigators